CLINICAL TRIAL: NCT06157216
Title: Circulating Tumor DNA Minimal Residual Disease-guided Adjuvant Chemotherapy in Patients With Stage II-III Gastric Cancer
Brief Title: Minimal Residual Disease-guided Adjuvant Therapy for Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Jinan Central Hospital (Other); Yantai Yuhuangding Hospital (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRD-GATE
Record Dates: First submitted 2023-11-19; First posted 2023-12-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Stage II-III Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD-guided treatment (Experimental): Patients post-surgery will receive MRD tests and receive MRD-guided adjuvant therapies. After that, MRD status will be continuously monitored for three years to guide the following therapies.
  Interventions: Drug: MRD-guided therapy

INTERVENTIONS:
Drug: MRD-guided therapy — MRD negative stage II gastric cancer: Observation; MRD negative stage III gastric cancer: S1 (40-60 mg, PO, bid, d1-d14 q3w); MRD positive stage II/III gastric cancer: XELOX (Oxaliplatin 130mg/m2, d1 +Capecitabine 1000mg/m2，PO. bid, d1-14, q3w) or SOX (Oxaliplatin 130mg/m2, d1 +S-1 40-60 mg, PO. bid, d1-14, q3w); MRD-negative patients will receive XELOX or SOX if MRD becomes positive.

SUMMARY:
This is a multicenter, single-arm, interventional study to explore the feasibility of circulating tumor DNA (ctDNA)-MRD testing to guide postoperative adjuvant treatment strategies in patients with stage II-III gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone D2 gastrectomy, achieved R0 resection, and are pathologically diagnosed with stage II-III gastric cancer.
2. No preoperative neoadjuvant or adjuvant therapy received.
3. Voluntary participation with signed informed consent, demonstrating good compliance and willingness to cooperate with follow-up procedures.
4. Age between 18-75 years, with no gender restrictions.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Estimated survival of 6 months or more.
7. Baseline hematological and biochemical parameters within specified limits: a. Hemoglobin ≥ 80g/L. b. Absolute neutrophil count ≥ 1.5×10^9/L. c. Platelet count ≥ 100×10^9/L. d. Aspartate or alanine aminotransferase ≤ 2.5 times the upper limit of normal. e. Alkaline phosphatase ≤ 2.5 times the upper limit of normal. f. Thyroid-stimulating hormone (TSH) ≤ 1 times the upper limit of normal (if abnormal, T3 and T4 levels must be normal).

Exclusion Criteria:

1. Pregnant or lactating women, or women of childbearing potential with a positive pregnancy test at baseline.
2. Evidence of postoperative recurrence or metastasis.
3. Previous anti-tumor therapy, including chemotherapy, radiotherapy, or immunotherapy.
4. Positive resection margins identified in postoperative pathology.
5. History of other malignancies within the past five years, except certain skin cancers, superficial bladder cancer, in situ cervical or breast cancer.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites.
7. Severe cardiovascular conditions such as symptomatic coronary artery disease, congestive heart failure (grade ≥ II), uncontrolled arrhythmias, or myocardial infarction within the last 12 months.
8. Uncontrolled infection, severe kidney disease, or other significant concurrent diseases.
9. Allergic reactions to study drugs.
10. Receipt of any anti-tumor therapy within 4 weeks prior to enrollment.
11. Administration of live attenuated vaccines within 4 weeks prior to the first study treatment dose or plans to receive such vaccines during the study period.
12. Positive HIV antibody, active hepatitis B or C (with specific viral load criteria).
13. Positive for COVID-19 nucleic acid or antigen test.
14. Other conditions deemed by the investigator to potentially affect patient safety or trial compliance, including serious illnesses requiring treatment, severe laboratory abnormalities, or other social or family reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-Free Survival (DFS) rate | 3-year after the last subject participating in
  The 3-year DFS rate is defined as the percentage of patients who remain free of tumor recurrence or death within three years after surgery.

SECONDARY OUTCOMES:
Rate of De-escalation Treatment | 3-year after the last subject participating in
  The Rate of De-escalation Treatment is defined as the proportion of patients among a study population who receive a reduction in the intensity or scope of therapeutic interventions.
Disease-Free Survival (DFS) | 3-year after the last subject participating in
  Disease-Free Survival (DFS) is defined as the duration of time from the initiation of surgery until the recurrence of the disease or death from any cause, whichever comes first.
Cumulative Risk of Recurrence | 3-year after the last subject participating in
  The Cumulative Risk of Recurrence is defined as the cumulative probability or risk of disease recurrence over a specified period, considering the entire study population.
3-year Overall Survival (OS) Rate | 3-year after the last subject participating in
  3-year Overall Survival (OS) Rate is defined as the percentage of patients who are still alive three years after the initiation of a specific treatment, regardless of disease recurrence or progression.

OTHER OUTCOMES:
Association between prognosis with multi-omic sequences | 3-year after the last subject participating in
  Association between prognosis with multi-omics data, including whole-exome sequencing, RNA sequencing, etc.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Qilu Hospital of Shandong Univertisy, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: Undecided